CLINICAL TRIAL: NCT03928808
Title: Safety and Efficacy of Fecal Microbiota Transplantation (FMT) in the Treatment of Severe and Enduring Anorexia Nervosa (SE-AN)
Brief Title: Fecal Microbiota Transplantation (FMT) in Treatment of Severe and Enduring Anorexia Nervosa
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Withdrawn due to covid-19 protocols on inpatient eating disorders unit.
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: OpenBiome (Industry); Foundation of Hope, North Carolina (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 18-1150
Record Dates: First submitted 2019-04-23; First posted 2019-04-26 (Actual); Last update posted 2023-01-30 (Actual); Status verified 2023-01

CONDITIONS: Anorexia Nervosa
Keywords: Fecal Microbiota Transplantation
MeSH Terms: conditions — Anorexia Nervosa | interventions — Fecal Microbiota Transplantation

STUDY DESIGN:
Intervention Model Description: Open Label Pilot Study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- FMT for SE-AN (Experimental): Inpatients at the UNC-Chapel Hill Center of Excellence for Eating Disorders (CEED) and will receive weekly fecal microbiota transplantations for four weeks. This will be in addition to standard care at CEED.
  Interventions: Biological: Fecal Microbiota Transplantation (FMT)

INTERVENTIONS:
Biological: Fecal Microbiota Transplantation (FMT) — Nasogastric administration of OpenBiome 25 g/mL solution administered nasogastrically once weekly for 4 consecutive weeks
  Other Names: OpenBiome FMT Upper Delivery formulation; FMP30

SUMMARY:
This is an open-label pilot study designed to explore the safety, feasibility, tolerability, and acceptability of fecal microbiota transplantation (FMT) in the treatment of severe and enduring anorexia nervosa (SE-AN).

DETAILED DESCRIPTION:
Open-label investigation of 10 individuals seeking inpatient treatment for severe and enduring anorexia nervosa. In addition to standard inpatient treatment, patients receive one FMT per week for 4 weeks, with follow-ups at 8 weeks and 6 months. Patients will receive 30 mL of healthy fecal microbial preparation (OpenBiome, FMP30) into the upper GI tract via a nasogastric tube weekly for 4 weeks. Primary outcomes are to determine safety, feasibility, tolerability, and acceptability of FMT for the treatment of AN. Secondary outcomes are: to determine preliminary efficacy as indexed by weight gain and weight retention over follow-up; to assess positive change in psychological metrics; to measure the efficiency of microbial transfer from the FMT material to the recipient intestinal microbiota; and to determine the duration of this effect via repeat stool sampling paired with 16S rRNA gene and/or shallow shotgun metagenomics.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated informed consent form.
* Stated willingness to comply with all study procedures and availability for the duration of the study.
* Female aged 18-45.
* Diagnosed with SE-AN, defined here as having suffered from AN for five or more years and having participated in two or more inpatient or residential treatment programs followed by weight relapse.
* Sufficiently medically stable to receive FMT (serum electrolytes within normal limits, normal EKG)
* Willing to adhere to the FMT dosing regimen.
* For females of reproductive potential, in sexual relationships with men, must use an acceptable method of contraception from 30 days prior to enrollment until 4 weeks after completing study treatment.* Participants must also be willing to be subjected to periodic pregnancy tests.
* Agreement to adhere to Lifestyle Considerations throughout study duration.
* Adequate insurance to cover inpatient stay.

  * Lifestyle Considerations: During this study, participants are asked to:

    * Participate in standard inpatient treatment at UNC-Chapel Hill's CEED.
    * Remain nil per os (npo) on the morning of each dosing session and for two hours after receiving FMT, on four individual instances of FMT administration.
    * Abstain from sexual activity or use a condom or other form of highly effective birth control during the 30-day active stage of the clinical trial.
    * Inform the research team as soon as possible if they become pregnant during the eight-week and six-month follow-up periods.
    * If a trial participant has begun a course of one of this trial's prohibited medications during the eight-week or six-month follow-up periods, participants will be asked only to report the name of the medication, dose, and duration of treatment.

Exclusion Criteria:

* Male or outside of the 18-45 range
* Previous FMT or microbiome-based products at any time excluding this study
* Patients with allergies to ingredients Generally Recognized As Safe (GRAS)
* Patients with a history of severe anaphylactic or anaphylactoid food allergy
* Patient received antibiotics in the last 48 hours. Patients will be eligible to enroll if antibiotic therapy is discontinued for at minimum 48 hours prior to start of study
* Requires continued antibiotic use or anticipates antibiotic use in the upcoming 4 weeks
* Concurrent intensive induction chemotherapy, radiation therapy, or biological treatment for active malignancy.
* Pregnancy or lactation
* Febrile illness within past month
* Treatment with another investigational drug within the past month
* Alcohol or drug dependence either at time of the study or within the last year
* Active gastrointestinal infection at time of enrollment
* Any gastrointestinal or potentially intestinal microbiota-related conditions, including: Severe gastroparesis (e.g., gastric pacemaker) and any history of gastrointestinal illness (including but not limited to inflammatory bowel disease, irritable bowel syndrome, celiac disease, any gastrointestinal cancer, etc.)
* Major gastrointestinal surgery (e.g. significant bowel resection) within 3 months before enrollment. This does not include appendectomy or cholecystectomy
* Type 1 or 2 diabetes mellitus
* Known or suspected toxic megacolon and/or known small bowel ileus
* History of total colectomy or bariatric surgery
* Solid organ transplant recipients less than or equal to 90 days posttransplant or on active treatment for rejection
* If at risk for CMV/EBV associated disease (at investigator's discretion, e.g. immunocompromised), negative IgG testing for cytomegalovirus (CMV) or Epstein-Barr Virus (EBV).
* Patients who are immunocompromised
* Unable or unwilling to comply with protocol requirements
* Expected life expectancy < 6 months
* A condition that would jeopardize the safety or rights of the subject, would make it unlikely for the subject to complete the study, or would confound the results of the study

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2023-04-01 (Estimated); Primary Completion 2024-03 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Proportion of Participants with Adverse Events (AEs) | Through day 30 (±3 days)
  Safety 1
Proportion of Participants with a Severe Adverse Event (SAE) | Through day 30 (±3 days)
  Safety 2
Number of Participants Recruited | 3 years
  Feasibility 1, Ability to Recruit 10 Participants with SE-AN
Number of Participants Able to Complete 4 FMT Administrations | 3 years
  Tolerability 1
Number of Participants Reporting Acceptable Levels of GI distress Post FMT | Through Week 4
  Tolerability 2

SECONDARY OUTCOMES:
Change in BMI Across Treatment and Follow-Up | Pre-Treatment through Follow-Up (Month 6)
  BMI calculated as weight in kg / height in meters squared
Change in Percent Body Fat Across Treatment and Follow-Up | Pre-Treatment through Follow-Up (Month 6)
  Body fat percentage (to the nearest 0.1%) will be measured using a Tanita Dual Frequency Total Body Composition Analyzer that assesses weight and bioelectrical impedance for adiposity.
Eating Disorder Examination Questionnaire (EDE-Q) Scores over Time | Pre-Treatment through Follow-Up (Month 6)
  The EDE-Q is a 28-item questionnaire measuring eating pathology and is derived directly from the Eating Disorder Examination Interview. The EDE-Q focuses on the past 28 days to assess the main behavioral (eating and purging) and attitudinal features of eating disorders. The 28 items are rated by the participant on a 7-point scale (ranging from 0 to 6), with higher scores indicating increased pathology. The EDE-Q includes 4 subscales: Restraint, Eating Concern, Weight Concern, and Shape Concern. The global score is the average of all 28 items, with a range of 0 to 6.
PHQ-9 Scores Over Time | Pre-Treatment through Follow-Up (Month 6)
  The Patient Health Questionnaire (PHQ-9) has 9 items with each rated from 0 to 3. Overall scores ranges from 0 to 27 with 1-4 being minimal depression, 5-9 being mild depression, 10-14 being moderate depression, 15-19 being moderately severe depression and 20-27 being severe depression.
GAD-7 Scores Over Time | Pre-Treatment through Follow-Up (Month 6)
  Anxiety symptoms as measured by the Generalized Anxiety Disorder (GAD-7) 7-item scale. The range of the measure is 0 to 21, with higher scores indicating greater anxiety symptoms.
PROMIS-GI Scores Over Time | Pre-Treatment through Follow-Up (Month 6)
  Self-reported outcome of GI symptom burden measured using the Patient-Reported Outcomes Measurement Information System (PROMIS) gastro-intestinal (GI) Symptoms scale on the study iPad. The scale includes 4 items and responses to each item are on a 1 (Never) to 5 (Almost Always) scale. Higher scores indicate greater GI symptom burden.

OTHER OUTCOMES:
FMT Transfer Efficiency | Pre-Treatment through Follow-Up (Month 6)
  The investigators will establish which particular taxa of bacteria from the FMT material successfully engrafted into the recipient's intestinal tract. FMT transfer efficiency is the percentage of bacterial taxa that successfully transfer from the donor FMT to the FMT recipient's stool.

CONTACTS AND LOCATIONS:
Overall Officials: Mary Kimmel, MD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- UNC Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual participant data (IPD) will be made available by controlled access. Qualified researchers with documented evidence of ethical approval and a clear research and statistical analysis plan will be given access through a secure file transfer protocol (FTP) site. Data to be shared include diagnostic information, age, non-identifying demographic data (including BMI and other anthropometric measures), psychometric, and sequence data along with a data dictionary.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 6 months after publication of the primary publication
Access Criteria: To qualified applicants with documented IRB approval and analytic plan. A Data Use Agreement must be executed with UNC prior to actual sharing of data.